CLINICAL TRIAL: NCT01699997
Title: The Use of Oxytocin as Adjunctive Therapy for the Treatment of Schizophrenia: a Randomized, Double Blind Trial
Brief Title: Oxytocin as Adjunctive Therapy for Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Giovanni de Girolamo, M.D., Responsible of Psychiatric Epidemiology and Evaluation Unit, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RF-2010-2311148
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Oxytocin; RCT
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): Each treatment will consist of 10 insufflations (5/nostril alternating between nostrils) of OXT Spray, which contains approximately 40 international units (IU) of OXT
  Interventions: Drug: Oxytocin
- Placebo vial (Placebo Comparator): Each treatment will consist of 10 insufflations (5/nostril alternating between nostrils) of placebo Spray, which contains all OXT Spray ingredients except for oxytocin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal spray with 40 IU of OXT
  Arms: Oxytocin
Drug: Placebo — Intranasal spray with placebo solution
  Arms: Placebo vial

SUMMARY:
Background: A large body of research has shown that Oxytocin (OXT) is an important prosocial peptide and there is also initial evidence that the central OXT system is altered in several mental disorders that are characterized by severe social disturbances and deficits, such as anxiety disorders with prominent social dysfunction (e.g., schizophrenia), mood disorders and borderline personality disorder. OXT may reduce psychotic symptoms and may diminish certain social cognition deficits that are not improved by current antipsychotic medications.

Aims: The project has two main aims, listed below:

1. To assess the efficacy of intranasal OXT in reducing negative symptoms in patients with schizophrenia in association with second-generation antipsychotics (SGA);
2. To use an Emotional Priming Paradigm task to assess pre- and post-treatment change in the patients general cognitive and emotional status.

Study Design: Randomized, double-blind, placebo-controlled, cross over design. Materials and methods: Patients involved in the study will be recruited in six centres in the north of Italy. Each subject (aged 18-45, with a duration of the disorder no longer than 10 years) will be enrolled after a screening phase. 80 patients will be randomly assigned to either 40 IU OXT once daily or vehicle placebo, in addition to their pre-study antipsychotic medication regimen: all reasonable attempts maintain the same SGA dosages throughout the study will be made. The study ratio is 1:1. The total study duration for each individual subject will be approximately 8 months, which includes an up to 7-day screening period, a baseline randomization visit, and a four month long cross-over treatment period. Subjects will be trained by researchers about the self-administration of intranasal OXT. A trustworthy caregiver will be trained as well. Each patient will receive every morning a SMS text message on his mobile phone as a reminder for OXT administration.

Before starting the treatment, all patients will be assessed with standardized assessment instruments and will undergo an in depth neuropsychological assessment; additional evaluations, including safety evaluations, will be performed at 4 and 8 month follow-ups.

The primary outcome measure will be the negative score in the Positive and Negative Syndrome Scale (PANSS) performed at 2,4,6 and 8 months since the start of the treatment.

DETAILED DESCRIPTION:
The project has two main aims:

1. Aims of the cross-over study To assess the efficacy of intranasal OXT in reducing negative symptoms in patients with SZ (as evaluated with PANSS), in association with standard Second Generation Antipsychotics (SGA)treatment; recruited patients will be aged 18-45 years and will have a disorder duration of no longer than 10 years.
2. Aims of the neuropsychological assessment To use an Emotional Priming Paradigm (EPP) task to assess pre- and post-treatment change in the patients general cognitive and emotional status.

The investigators aim at treating a large sample size of patients with schizophrenia, consisting exclusively of patients with a limited disorder duration and rather young age, for a sufficiently long period of time. Our rationale for employing a longer treatment period than used in previous and on-going trials is to ascertain the possibility of a positive OXT dose-response relationship, which would be observable, however, with longer treatment exposure. Moreover, only patients with a disorder onset of 10 years or less will be enrolled.

They will then be standardized in terms of AP treatment and randomized to OXT or placebo for 8 months.

OXT is a hormone that is naturally present in the human body, and recent studies have suggested that patients with SZ show low levels of this neuropeptide. It is therefore hypothesized that the treatment proposed in this project might balance apparently lower OXT levels in these patients.

Finally, another innovative aspect of this project is the attention at ameliorating patients adherence to treatment by supporting them with a reminder program (automatic SMS will be sent every morning to remind patients the daily OXT self-administration) and involving a trustworthy caregiver who will be trained in OXT administration and will be asked to monitor the patient compliance by recording each self-administration on a written form.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of SZ, according to DSM-IV criteria, for at least one year, evaluated with SCID/P
* A minimum PANSS total score of 55 (indicating moderate severity, due to ongoing AP treatment) .
* A minimum CGI-S score of 4
* Age between 18 and 45 years
* A disorder duration of no longer than 10 years
* Women of childbearing age must test negative for pregnancy at the time of enrolment.

All patients must:

* be on a therapeutic dose of a SGA (or a maximum 2 SGAs) with no major dose changes for at least 4 weeks.
* have the ability to provide informed consent
* be able to use a nasal spray
* reside in the service catchment area
* show evidence of no alcohol or substance dependence in the last year

Exclusion Criteria:

* Diagnosis of mental retardation
* Diagnosis of organic mental disorder
* History of no response to treatment with clozapine
* History of hypersensitivity to OXT or vehicle
* Alcohol or substance dependence in the last year
* Presence of, or history of clinically significant allergic rhinitis as assessed by the treating clinician
* Being pregnant or breastfeeding
* Having given birth in the past 6 months or breast-feeding in the past 3 months
* Low literacy as indicated by an inability to read and understand the consent form

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in PANSS negative score, as measured at T0 and at 2,4,6 and 8 months. | 8 months
  Using the PANSS negative score as primary end-point, the investigators expect to observe a reduction in PANSS negative subscale scores in the treated group ranging from 0.9 to 2, with an effect size Cohens d=0.45, in agreement with the results of a previous study, in which authors who observed a reduction of 1.7 with an effect size Cohens d= 0.5. The investigators also expect that OXT will have a positive influence on the patients quality of life and reduction of PANSS positive subscale score. Correlations between OXT plasma levels, symptoms, and response to treatment will be evaluated to identify respondent and non-respondent patient groups

SECONDARY OUTCOMES:
PANSS total score change. | 8 months
  The secondary end-point will be the PANSS total score

OTHER OUTCOMES:
Brief Assessment of Cognitive deficits in Schizophrenics (BACS) score change | 8 months
Reading the Mind in the Eyes Test (RMET) score change. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Girolamo, M.D., Principal Investigator — IRCCS Fatebenefratelli, Brescia
Locations (7):
- Italy (7):
  - Statistical Unit, Institute of Biomathematics, University of Urbino, Urbino, Pesaro Urbino
  - IRCCS Fatebenefratelli, Brescia
  - Department of Mental Health, Desenzano
  - Institute of Neuroscience, National Research Council, Milan
  - Department of Mental Health, Padua
  - Psychiatric Clinic, University of Pisa, Pisa
  - Psychiatric Clinic, University of Udine, Udine

REFERENCES:
- [Derived] Dagani J, Sisti D, Abelli M, Di Paolo L, Pini S, Raimondi S, Rocchi MB, Saviotti FM, Scocco P, Totaro S, Balestrieri M, de Girolamo G. Do we need oxytocin to treat schizophrenia? A randomized clinical trial. Schizophr Res. 2016 Apr;172(1-3):158-64. doi: 10.1016/j.schres.2016.02.011. Epub 2016 Feb 14. PMID 26883950
- [Derived] Lee MR, Wehring HJ, McMahon RP, Liu F, Linthicum J, Verbalis JG, Buchanan RW, Strauss GP, Rubin LH, Kelly DL. Relationship of plasma oxytocin levels to baseline symptoms and symptom changes during three weeks of daily oxytocin administration in people with schizophrenia. Schizophr Res. 2016 Apr;172(1-3):165-8. doi: 10.1016/j.schres.2016.02.014. Epub 2016 Feb 12. PMID 26879587
- See also: This is the website of the Coordinating Centre — http://www.irccs-fatebenefratelli.it/